CLINICAL TRIAL: NCT06805500
Title: Robotic Assisted Balance and Exoskeleton Training (REACTION) in Neurorehabilitation: a Feasibility Study
Acronym: REACTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roessingh Research and Development (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL 2025-17884; 1789 (Other Grant/Funding Number: EUREKA)
Record Dates: First submitted 2025-01-16; First posted 2025-02-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Spinal Cord Injury
Keywords: exoskeleton; gait trainer; neurological disease; rehabilitation
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Multicentred feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Device: REACTION; Device: ABLE Regain; Device: GABLE Core

INTERVENTIONS:
Device: REACTION — Combination of a exoskeleton and gait trainer
Device: ABLE Regain — Exoskeleton
Device: GABLE Core — Gait trainer

SUMMARY:
The goal of this clinical trial is to explore the effect on walking speed of a new robotic assisted balance and gait trainer (REACTION) and their subsystems in individuals with neurological disorders. The study will provide insight in the feasibility of REACTION.

Participants will:

* Participate in two sessions in which every session contains a walking task and balance tasks
* end the study with a semi-structured interview

DETAILED DESCRIPTION:
The first day will be focusing on 4 conditions: tasks without aid, tasks with regular aid, task with the ABLE Regain and tasks with REACTION. The first and third condition consist of a walking task and balance tasks, The second and fourth condition is only focusing on the walking task with the aim of getting familiar to the device and the walking task.

The second day will also be focusing on four conditions: tasks without aid, tasks with aid, tasks with the GABLE Core and task with REACTION (Fig 3.2). The conditions 'tasks without aid', 'tasks with the GABLE Core' and 'tasks with REACTION' consist of a walking task and balance tasks (similar to day 1). The condition 'tasks with aid' only consists of a walking task.

A semi-structured interview with the corresponding physiotherapist and patient will be held to gather more information about usability and feasibility of REACTION from a therapist's and patient's perspective.

ELIGIBILITY:
In order to be eligible to participate in this study, a participant must meet all of the following criteria:

* Age > 16 years
* Able to give informed consent

Stroke patients:

* first-ever ischemic or haemorrhagic stroke
* FAC score between 3 and 4
* (Sub)acute or chronic phase

SCI patients:

* Neurological injury levels ranging from C5 to T9
* Motor incomplete spinal cord injury (ASIA impairment score of C or D)
* Able to walk independently (without physical support)

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study:

* Premorbid disability of lower extremity
* Progressive neurological diseases like dementia or Parkinson
* Skin lesions or severely impaired sensation at the hemiparetic leg
* Contraindication for mobilization, like lower limb fracture
* Insufficient knowledge of the Dutch language to understand the purpose or meth-ods of the study
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Walking speed | 1 week
  The walking speed of the participants during a 6.5 meter walk.

SECONDARY OUTCOMES:
Kinematic data | 1 week
  Kinematic data, such as the joint angles, will be measured with IMUs
Short Form Berg Balance Scale (SFBBS) | 1 week
  The balance will be assessed with the Short Form Berg Balance Scale (SFBBS). SFBBS consists of a 7-items scale that measures static and dynamic balance. Each item has a 3-point score (0, 2 and 4 from original Berg Balance Scale). Total score ranges from 0 (poor balance) to 28 (good balance).
DON/DOFF | 1 week
  The time to put the device on (DON) and the device off (DOFF)
Level of Assistance | 1 week
  The level of assistance will be assessed based on the settings of the device

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Roessingh Research and Development, Enschede
  - Sint Maartenskliniek, Ubbergen

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request